CLINICAL TRIAL: NCT05482763
Title: Pilot Study on the Evaluation of the Efficacy, Tolerability and Safety of Topical and Oral Antifungals in the Treatment of Onychomycosis and Creation of a Library of Dermatological Clinical Isolates
Brief Title: Mycosis Culture Collection From Dermatological Isolated
Acronym: MYCDERM
Status: Active, not recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Elena Campione, Principal Investigator, University of Rome Tor Vergata
Other Study IDs: N. 143.22
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Onychomycosis; Resistant Infection; Nail Diseases
Keywords: Onychomycosis; Resistant Infection; Nail Diseases
MeSH Terms: conditions — Onychomycosis; Nail Diseases | interventions — Itraconazole; Terbinafine; amorolfine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Nail
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with onychomycosis: All patients with clinical suspicion of onychomycosis at the Tor Vergata Polyclinic center will be enrolled according to the inclusion and exclusion criteria of the study. After signing the informed consent, the subjects will be subjected to scraping or clipping of the nail unit affected by the disease. The collected material will be stored in a sterile container to be sent to the Microbiology laboratory.
  Interventions: Drug: Terbinafine Topical Gel; Drug: Itraconazole 200 mg; Drug: Terbinafine 250 mg; Drug: Ciclopirox Topical Gel; Drug: Amorolfine 50 MG/ML

INTERVENTIONS:
Drug: Terbinafine Topical Gel — Topical application of terbinafine
Drug: Itraconazole 200 mg — systemic itraconazole pulse therapy
Drug: Terbinafine 250 mg — systemic terbinafine
Drug: Ciclopirox Topical Gel — Topical application of ciclopirox
Drug: Amorolfine 50 MG/ML — Topical application of amorolfine

SUMMARY:
This pilot, prospective, observational drug study aims to evaluate the efficacy, tolerability and safety of topical and oral antifungals in the treatment of onychomycosis caused by yeasts, dermatophytic moulds and non-dermatophytic moulds as well as correlate the scores in the MALDI-TOF method for the 'identification of genus and species of higher fungi utilizing the comparison between identification in direct optical microscopy, culture examination and optical microscopy and macroscopic and onychoscopic clinical aspects. Furthermore, an optional substudy will evaluate the drug resistance of clinical isolates using molecular or genetic methods.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical suspicion of onychomycosis.

Exclusion Criteria:

* Patients deemed unsuitable by the investigator
* Patients with documented sensitivity to study drugs such as azoles, allylamine, and ciclopirox olamine.
* Failure to adhere to topical or oral therapy;
* Replacement of the therapy reported in the study protocol;
* Voluntary decision by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study involves the collection of biological material from patients with clinical suspicion of onychomycosis at an initial time, baseline T0, prior to the first administration of therapy according to the Italian guidelines, and evaluation with follow-up visits at 3,6,9 and 12 months of treatment (T3-T12).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Change of Onychomycosis Severity Index (OSI) | week 0,12,24,36,52
  Change of Onychomycosis Severity Index (OSI) from baseline to 12 months:
  * Area of Involvement (0-5 points)
  * Proximity of Disease to Matrix (1-5 points)
  * Presence of Dermatophytoma or Subungual Hyperkeratosis 2 mm ( 0 or 10 points)
Safety and Tolerability: Established from patient incidence of Treatment-Emergent Adverse Events | Monitored from screening visit to end of study visit (52 week)
  Indicated by the number of patients with treatment-related adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE).
Complete Cure at 12 months in the Target Toes | Week 52
  Complete Cure is defined as 1) 100% healthy, clear nail, and 2) negative mycology. Healthy, clear nail is absent any disease involvement attributable to DLSO and is determined by Investigator Global Assessment (IGA). Negative mycology is defined as zero visualization of septate hyphae by KOH microscopy (negative KOH) combined with a fungal culture negative for causal dermatophytes (negative fungal culture).

SECONDARY OUTCOMES:
Change in Dermatology life Quality Index (DLQI) | week 0,12,24,36,52
  Evaluation of the quality of life of treated patients before and after treatment (0-30 points)
Patient Global Assessment | week 0,12,24,36,52
  To establish each patient's impression of DLSO improvement in their target toe over the study period, patients will reference the following scale (0 = clear of DLSO, 1 = marked improvement of DLSO, 2 = moderately improved DLSO, 3 = slightly improved DLSO, 4 = unchanged, 5 = worse)

OTHER OUTCOMES:
Rate of correct classification by the test (MALDI-TOF MS profiling) from positive cultures | Week 0
  For each culture positive clinical sample, the status ("correct" or "incorrect") of the classification of the sample ("infected" or "not infected") by the test (MALDI-TOF MS profiling) will be determined. Then the rate of correct classification will be calculated. The test will be considered efficient when it has reached a correct classification rate of more than 95%.
Rate of correct classification by KOH Test from clinical isolates | Week 0
  For each clinical sample, the status ("correct" or "incorrect") of the classification of the sample ("infected" or "not infected") by the KOH test will be determined. Then the rate of correct classification will be calculated. The test will be considered efficient when it has reached a correct classification rate of more than 95%.
Rate of correct classification by direct Microscopy Test from positive cultures | Week 0
  For each culture positive clinical sample, the status ("correct" or "incorrect") of the classification of the sample ("infected" or "not infected") by the test (Microscopy of the cultures) will be determined. Then the rate of correct classification will be calculated. The test will be considered efficient when it has reached a correct classification rate of more than 95%.
Correlation between the identified fungi pathogens and the clinical course of the participants. | Week 52
  In fungi infected participants, the presence of a correlation between the presence of fungal infection and the clinical evolution of patients will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Campione, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- Tor Vergata Univerisity Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No